CLINICAL TRIAL: NCT06591117
Title: A Prospective, Multicenter Clinical Study to Evaluate the Safety and Efficacy of the Vizio Aqueous Microshunt for the Treatment of Refractory Glaucoma
Brief Title: Vizio Aqueous Microshunt Clinical Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ocumedex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C100
Record Dates: First submitted 2024-08-14; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Refractory Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: Vizio Aqueous Microshunt (VAM) - an implantable device intended to reduce intraocular pressure (IOP) by shunting aqueous humor from the anterior chamber to the surface of the eye.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vizio Treatment (Experimental): single-arm clinical study
  Interventions: Device: Vizio Aqueous Microshunt

INTERVENTIONS:
Device: Vizio Aqueous Microshunt — Ocular microshunt placement for the treatment of Glaucoma

SUMMARY:
Evaluate the Safety and Efficacy of the Vizio Aqueous Microshunt for the Treatment of Refractory Glaucoma

DETAILED DESCRIPTION:
A Prospective, Multicenter Clinical Study to Evaluate the Safety and Efficacy of the Vizio Aqueous Microshunt for the Treatment of Refractory Glaucoma

ELIGIBILITY:
Inclusion Criteria:

1. Age 22-85 years.
2. Refractory glaucoma describes eyes uncontrolled by medical therapy and diagnosed with glaucoma which meet at least one of the following criteria: 1) Failed one or more incisional intraocular glaucoma surgeries (e.g., glaucoma filtering surgery or tube shunt); 2) Failed one or more cilioablative procedures (e.g., cryotherapy, cyclodiode therapy); 3) Have any other condition (e.g., conjunctival scarring, uveitis) in which a conventional incisional glaucoma surgery like trabeculectomy would be more likely to fail than for an eye with uncomplicated primary open angle glaucoma.
3. Primary open-angle or traumatic glaucoma.
4. Medicated DIOP ≥25 mmHg and ≤45 mmHg on maximum-tolerated medical therapy that is stable for at least 30 days.
5. Best-corrected baseline visual acuity of light perception or better in study eye.
6. Glaucomatous optic nerve damage as evidenced by any of the following optic disc or retinal nerve fiber layer structural abnormalities:

   * Diffuse thinning, focal narrowing, or notching of the optic disc rim, especially at the inferior or superior poles with or without disc hemorrhage;
   * Localized abnormalities of the peripapillary retinal nerve fiber layer, especially at the inferior or superior poles; or
   * Optic disc neural rim asymmetry of the two eyes consistent with loss of neural tissue
7. Visual field mean deviation (MD) by Humphrey Visual Field: Visual field defects consistent with glaucomatous optic nerve damage and mean deviation worse than -3 dB in the study eye; and at least one of the following two findings:

   * A cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level on the pattern deviation (PD) plot;
   * Glaucoma hemi-field test "outside normal limits."
8. At least two contiguous clock hours of intact conjunctiva near the limbus between clock hours of 10:00 and 02:00 in the study eye.
9. Adequate space in the anterior chamber by Spaeth Grade C, D or E for iris insertion (with indentation).
10. Participant has the understanding, ability, and willingness to fully comply with study procedures and postoperative care instructions.
11. Participant understands, is capable and competent to sign the informed consent.

Exclusion Criteria:

1. Active neovascular conditions such as active iris or corneal neovascularization, or active proliferative retinopathy in study eye.
2. Pigmentary glaucoma in study eye.
3. Pseudoexfoliation syndrome in study eye.
4. Angle-closure glaucoma in study eye.
5. Iridocorneal endothelial syndrome in study eye.
6. Uveitic glaucoma in the study eye.
7. Epithelial or fibrous downgrowth in the study eye.
8. Corneal conditions in study eye inhibiting normal incisional healing (e.g. Fuch's dystrophy) or would impair visualization of implant inside anterior chamber.
9. Prior intraocular surgery in study eye within ≤6 months before the preoperative visit (including phacoemulsification).
10. Central corneal endothelial cell count of less than 1600 cells/mm2 in the study eye.
11. Anticipated need for ocular surgery or retinal laser procedure in the study eye within the 12-month follow-up period.
12. Need for glaucoma surgery combined with other ocular procedures in the study eye at time of implant (e.g. cataract surgery, penetrating keratoplasty, or retinal surgery).
13. Unwilling to discontinue contact lens use in the study eye after surgery.
14. Central corneal thickness ≤490μm or ≥620μm.
15. Clinically significant inflammation or infection in the study eye within 60 days prior to the preoperative visit (e.g., blepharitis, conjunctivitis, keratitis, uveitis, herpes simplex infection) or any systemic infection. For purposes of this study, clinically significant is considered any such condition requiring prescription therapy.
16. Any condition that prevents the device implantation in the superior region of the study eye.
17. Vitreous in the anterior chamber for which a vitrectomy is anticipated.
18. Functionally significant cataract in the study eye.
19. Other clinical conditions:

    1. Poorly controlled diabetes (Type I or Type II) as determined by HbA1c >8 within 3 months of implant.
    2. Cancer requiring treatment during the duration of the study.
    3. Any drugs (e.g.: immunosuppressive drugs) or co-morbidity that might inhibit wound healing.
20. Participation in any other clinical study during participation in this study.
21. Engage in activities that involve submerging their head under water, such as diving or swimming.
22. Women who are (i) pregnant, (ii) nursing, (iii) planning a pregnancy and (iv) of childbearing potential not using a reliable method of contraception.
23. Life expectancy <1 year.

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 12 months
  The primary endpoint is a binary measure of at least 20% reduction from baseline in diurnal IOP at twelve monthsbaseline, on the same number or fewer topical IOP-lowering medications, based on intent-to-treat population.
Safety | 12 months
  Rate of occurrence of serious procedure-related and/or device-related adverse events at 12 months post implantation.

SECONDARY OUTCOMES:
Responder Rate | 12 months
  Responder rate for complete success at 12M: Defined as at least 20% mean diurnal IOP reduction from baseline after device implant with no IOP lowering medications
Overall Safety | 12 months
  Rate of all ocular and non-ocular adverse events (intraoperative complications and postoperative events), including rate of pre-specified ocular adverse events (per ANSI Z80.27) and abnormal findings by pachymetry, slit lamp biomicroscopy, gonioscopy, fundoscopy, specular microscopy and patient-reported symptoms